CLINICAL TRIAL: NCT01020747
Title: A Pilot Study to Evaluate the Effects of Antiangiogenic Factor as an Adjunct Treatment After Photoangiolysis in Patients With Bilateral Recurrent Respiratory Papillomatosis of the Vocal Fold
Brief Title: Bevacizumab for Treatment of Recurrent Respiratory Papillomatosis (RRP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven M. Zeitels, MD, FACS, Director: Center for Laryngeal Surgery and Voice Rehabilitation, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC-P001
Record Dates: First submitted 2009-11-13; First posted 2009-11-25 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2012-12-20 (Estimated); Status verified 2012-12

CONDITIONS: Recurrent Respiratory Papillomatosis
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — Bevacizumab; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Avastin® (bevacizumab) — Bevacizumab injections (~7.5-12.5mg in 0.3 - 0.5 c.c.) into diseased vocal folds in conjunction with 532 nm pulsed-KTP laser photoangiolysis, administered every 6 ±1 weeks, for a total of 5 treatments. No patient will have an injection volume exceed 0.5 cc. for any single treatment. If initial results indicate a benefit, as described below, an extension of the active treatment period will be permitted up to a total treatment duration of 18 months.
  Other Names: Avastin®
Drug: Saline — A sham injection with saline (0.3-0.5 cc) has been administered to the other vocal fold as the control. This therapy will be administered once every 6 ± 1 week for 6 months, with the same vocal fold selected for the initial treatment always getting the drug injection.

SUMMARY:
This phase I single center open labeled study is planned to assess the safety and tolerability of bevacizumab for treating patients with bilateral Recurrent Respiratory Papillomatosis (RRP). Approximately 20 patients will receive bevacizumab directly injected into the vocal folds. Patients who enroll in the protocol will be injected with bevacizumab in one vocal fold that represents the more diseased of the two folds. A sham injection with saline will be administered to the other vocal fold as the control. This therapy will be administered once every 6 ± 1 week for 6 months, with the same vocal fold selected for the initial treatment always getting the drug injection. The investigator will also treat lesions by laser photoangiolysis of both vocal folds using the 532 nm potassium-titanyl-phosphate (KTP) laser.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with dysphonia that have been diagnosed with Recurrent Respiratory Papillomatosis (RRP) of the vocal folds
* Age between 18 and 60 years old
* Female patients must be surgically sterilized, postmenopausal, or employ adequate contraception. Criteria for menopause are surgical menopause (hysterectomy, oophorectomy) or age > 45 years with absence of menses for greater than 12 months and an elevated serum Hormone, follicle-stimulating (FSH) (> 25 mIU/mL). Tubal ligation with menses within the past 12 months is not considered to be surgical sterilization.
* Have bilateral glottal papillomatosis (i.e., involving both the right and left vocal folds)
* Willing and able to comply with the investigational nature of the study and able to communicate well with investigators.
* Ability to comprehend and willingness to provide written informed consent in accordance with institutional and regulatory guidelines.

Exclusion Criteria:

* Have known sensitivity to bevacizumab
* Have been treated systemically with bevacizumab within 4 months (approximately 6 half-lives).
* Have hematocrits < 30, elevated PT or PTT levels more than 1.2 X the upper limit of normal (ULN) or absolute platelet counts below the lower limit of normal (LLN).
* Have absolute neutrophil counts below 1500
* Have urine dipsticks positive for ≥3+ proteinuria will have spot urine collections and those patients with urine protein to urine creatinine ratios greater than 1.5.
* Have a history of congestive heart failure, angina that remains symptomatic despite medications, myocardial infarction or coronary artery disease-related procedure within the past 6 months (including angioplasty, stent placement, bypass graft surgery) or who have prosthetic heart valves.
* Have significant uncontrolled hypertension (systolic blood pressure above 160 and/or diastolic blood pressure above 100).
* Have had surgeries within 1 month of enrollment or who have un-healed surgical incisions at screening.
* Have a history of thromboembolic events, gastro-intestinal (GI) ulcer or bleeding, or with a history of wound dehiscence.
* Female patients that are pregnant, nursing or plan to nurse during the up to 18 months of treatment period.
* Patients with a history of bleeding disorders, documented platelet dysfunction, current use of anti-platelet drugs, or abnormal prothrombin time (PT) or activated partial thromboplastin timea (PTT) laboratory values as defined in number 3 above.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Zeitels, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Anderson RR, Parrish JA. Selective photothermolysis: precise microsurgery by selective absorption of pulsed radiation. Science. 1983 Apr 29;220(4596):524-7. doi: 10.1126/science.6836297.
- [Background] Armstrong LR, Derkay CS, Reeves WC. Initial results from the national registry for juvenile-onset recurrent respiratory papillomatosis. RRP Task Force. Arch Otolaryngol Head Neck Surg. 1999 Jul;125(7):743-8. doi: 10.1001/archotol.125.7.743. PMID 10406310
- [Background] Avery RL, Pieramici DJ, Rabena MD, Castellarin AA, Nasir MA, Giust MJ. Intravitreal bevacizumab (Avastin) for neovascular age-related macular degeneration. Ophthalmology. 2006 Mar;113(3):363-372.e5. doi: 10.1016/j.ophtha.2005.11.019. Epub 2006 Feb 3. PMID 16458968
- [Background] Burns JA, Zeitels SM, Akst LM, Broadhurst MS, Hillman RE, Anderson R. 532 nm pulsed potassium-titanyl-phosphate laser treatment of laryngeal papillomatosis under general anesthesia. Laryngoscope. 2007 Aug;117(8):1500-4. doi: 10.1097/MLG.0b013e318064e869. PMID 17585283
- [Background] Dedo HH, Yu KC. CO(2) laser treatment in 244 patients with respiratory papillomas. Laryngoscope. 2001 Sep;111(9):1639-44. doi: 10.1097/00005537-200109000-00028. PMID 11568620
- [Background] Derkay CS. Task force on recurrent respiratory papillomas. A preliminary report. Arch Otolaryngol Head Neck Surg. 1995 Dec;121(12):1386-91. doi: 10.1001/archotol.1995.01890120044008. PMID 7488368
- [Background] Folkman J. Angiogenesis. Annu Rev Med. 2006;57:1-18. doi: 10.1146/annurev.med.57.121304.131306. PMID 16409133
- [Background] Franco RA Jr, Zeitels SM, Farinelli WA, Anderson RR. 585-nm pulsed dye laser treatment of glottal papillomatosis. Ann Otol Rhinol Laryngol. 2002 Jun;111(6):486-92. doi: 10.1177/000348940211100603. PMID 12090703
- [Background] Fung AE, Rosenfeld PJ, Reichel E. The International Intravitreal Bevacizumab Safety Survey: using the internet to assess drug safety worldwide. Br J Ophthalmol. 2006 Nov;90(11):1344-9. doi: 10.1136/bjo.2006.099598. Epub 2006 Jul 19. PMID 16854824
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Kernt M, Neubauer AS, Kampik A. Intravitreal bevacizumab (Avastin) treatment is safe in terms of intraocular and blood pressure. Acta Ophthalmol Scand. 2007 Feb;85(1):119-20. doi: 10.1111/j.1600-0420.2006.00819.x. No abstract available. PMID 17244226
- [Background] Meert AP, Feoli F, Martin B, Ninane V, Sculier JP. Angiogenesis in preinvasive, early invasive bronchial lesions and micropapillomatosis and correlation with EGFR expression. Histopathology. 2007 Feb;50(3):311-7. doi: 10.1111/j.1365-2559.2007.02610.x. PMID 17257126
- [Background] Mounts P, Shah KV, Kashima H. Viral etiology of juvenile- and adult-onset squamous papilloma of the larynx. Proc Natl Acad Sci U S A. 1982 Sep;79(17):5425-9. doi: 10.1073/pnas.79.17.5425. PMID 6291043
- [Background] Parsons DS, Bothwell MR. Powered instrument papilloma excision: an alternative to laser therapy for recurrent respiratory papilloma. Laryngoscope. 2001 Aug;111(8):1494-6. doi: 10.1097/00005537-200108000-00030. No abstract available. PMID 11568590
- [Background] Rahbar R, Vargas SO, Folkman J, McGill TJ, Healy GB, Tan X, Brown LF. Role of vascular endothelial growth factor-A in recurrent respiratory papillomatosis. Ann Otol Rhinol Laryngol. 2005 Apr;114(4):289-95. doi: 10.1177/000348940511400407. PMID 15895784
- [Background] Ratner M. Genentech discloses safety concerns over Avastin. Nat Biotechnol. 2004 Oct;22(10):1198. doi: 10.1038/nbt1004-1198. No abstract available. PMID 15470443
- [Background] Sachdev JC, Jahanzeb M. Evolution of bevacizumab-based therapy in the management of breast cancer. Clin Breast Cancer. 2008 Oct;8(5):402-10. doi: 10.3816/CBC.2008.n.048. PMID 18952553
- [Background] Shehab N, Sweet BV, Hogikyan ND. Cidofovir for the treatment of recurrent respiratory papillomatosis: a review of the literature. Pharmacotherapy. 2005 Jul;25(7):977-89. doi: 10.1592/phco.2005.25.7.977. PMID 16006276
- [Background] Spaide RF, Laud K, Fine HF, Klancnik JM Jr, Meyerle CB, Yannuzzi LA, Sorenson J, Slakter J, Fisher YL, Cooney MJ. Intravitreal bevacizumab treatment of choroidal neovascularization secondary to age-related macular degeneration. Retina. 2006 Apr;26(4):383-90. doi: 10.1097/01.iae.0000238561.99283.0e. PMID 16603955
- [Background] Steinberg BM, DiLorenzo TP. A possible role for human papillomaviruses in head and neck cancer. Cancer Metastasis Rev. 1996 Mar;15(1):91-112. doi: 10.1007/BF00049489. PMID 8842481
- [Background] Strong MS, Vaughan CW, Cooperband SR, Healy GB, Clemente MA. Recurrent respiratory papillomatosis: management with the CO2 laser. Ann Otol Rhinol Laryngol. 1976 Jul-Aug;85(4 Pt 1):508-16. doi: 10.1177/000348947608500412. PMID 949157
- [Background] Wu L, Martinez-Castellanos MA, Quiroz-Mercado H, Arevalo JF, Berrocal MH, Farah ME, Maia M, Roca JA, Rodriguez FJ; Pan American Collaborative Retina Group (PACORES). Twelve-month safety of intravitreal injections of bevacizumab (Avastin): results of the Pan-American Collaborative Retina Study Group (PACORES). Graefes Arch Clin Exp Ophthalmol. 2008 Jan;246(1):81-7. doi: 10.1007/s00417-007-0660-z. Epub 2007 Aug 3. PMID 17674014
- [Background] Zeitels, S.M. (2001). In Atlas of Phonomicrosurgery and Other Endolaryngeal Procedures for Benign and Malignant Disease (San Diego).
- See also: Avastin package insert and information from the Genentech website. — http://www.gene.com/gene/products/information/oncology/avastin
- See also: International RRP ISA site — http://www.rrpwebsite.org/
- See also: RRP Foundation website — http://www.rrpf.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Group Avastin: Subjects received Avastin in the more diseased vocal fold and saline in the other.
Period: Overall Study
Arm/Group | Group Avastin
Started | 20
Completed | 19
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Group Avastin
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: The Primary Activity Variable Was the Recurrence of Recurrent Respiratory Papillomatosis (RRP) in Bevacizumab Treated and the Un-treated Vocal Fold in the Same Patient During and at the End of the 6-month Treatment Period.
Description: Prior to each treatment,the area of reappearance of disease was measured and the % change from baseline was calculated. The change was then added to the % change from the previous treatment to generate a cumulative total % change of reappearance of RRP from baseline. The additive nature of this parameter resulted in % greater than 100% if the area of vocal fold affected by the RRP increased over the baseline measurement.
Time Frame: 6 months
Population: All subjects were analyzed.
Measure: Mean (Standard Deviation); unit: total percentage change
Groups:
- Bevacizumab Treated Vocal Fold: Subjects received injections of bevacizumab in conjunction with Potassium-Titanyl-Phosphate (KTP)laser photoangiolysis in the more diseased vocal fold.
- Untreated Vocal Fold: Subjects received saline injections in combination with Potassium-Titanyl-Phosphate (KTP)laser photoangiolysis in the less diseased vocal fold.
Arm/Group | Bevacizumab Treated Vocal Fold | Untreated Vocal Fold
Number analyzed (Participants) | 20 | 20
total percentage change | 85.3 (68.6) | 225.3 (191.1)

ADVERSE EVENTS:
Time Frame: The main treatment period lasted 6 months for each subject. Adverse events were captured for all subjects for a period of 26 months.
Arm/Group | Group Avastin
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 20/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group Avastin (N=20)
Aguesia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cold (Respiratory, thoracic and mediastinal disorders) | 1 (1)
cough/URI (Respiratory, thoracic and mediastinal disorders) | 1 (1)
disk herniation (Musculoskeletal and connective tissue disorders) | 1 (1)
Diminished voice volume (Respiratory, thoracic and mediastinal disorders) | 1 (1)
drainage and congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
dysphagia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
eye twitching (Eye disorders) | 1 (1)
flu-like symptoms (Infections and infestations) | 1 (1)
headache (General disorders) | 2 (2)
higher pitch (Respiratory, thoracic and mediastinal disorders) | 1 (1)
hoarseness (Respiratory, thoracic and mediastinal disorders) | 20 (20)
oversedation (Injury, poisoning and procedural complications) | 1 (1)
poison ivy rash (Skin and subcutaneous tissue disorders) | 1 (1)
toe (right) cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
tongue numbness (Injury, poisoning and procedural complications) | 2 (2)
tooth ache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No